CLINICAL TRIAL: NCT02837848
Title: Effect of Adding Muscle Coactivation to Regular Shoulder Strengthening Exercises on Function and Pain With Patients Suffering of Rotator Cuff Tendinopathy: A Single-Blind Randomized Controlled Trial
Brief Title: Effect of Muscle Coactivation Strengthening for Rotator Cuff Tendinopathy
Acronym: coacticuff
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Nathaly Gaudreault, Professor, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-1404
Record Dates: First submitted 2016-07-12; First posted 2016-07-20 (Estimated); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Tendinopathy
Keywords: Rotator Cuff Tendinopathy; Exercises; Coactivation; Strengthening
MeSH Terms: conditions — Tendinopathy; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Coactivation strengthening (Experimental): Coactivation strengthening implies a recruitment of the pectoralis major and the latissimus dorsi while performing regular strengthening.
  Interventions: Procedure: Coactivation Strengthening
- Regular strengthening (Active Comparator): Regular strengthening implies external rotation, internal rotation, flexion and abduction of the gleno-humeral joint and scapular protraction and retraction of the scapulothoracic joint strengthening.
  Interventions: Procedure: Regular Strengthening

INTERVENTIONS:
Procedure: Coactivation Strengthening — Coactivation strengthening implies a recruitment of the pectoralis major and the latissimus dorsi while performing regular strengthening.
  Arms: Coactivation strengthening
Procedure: Regular Strengthening — Regular strengthening implies external rotation, internal rotation, flexion and abduction of the gleno-humeral joint and scapular protraction and retraction of the scapulothoracic joint strengthening.
  Arms: Regular strengthening

SUMMARY:
Rotator cuff tendinopathy (RCT) is the most frequent cause of shoulder pain. RCT is frequently termed as impingement syndrome, based on the underlying mechanism in which the subacromial space soft tissues (subacromial bursa, rotator cuff tendons and long head of the biceps tendon) get encroached under the coracoacromial arch when the arm is elevated. RCT contributes in the decrease in quality of life and function, and in inducing work incapacities and sleep disorders.

Exercises, as conservative management, were shown to be effective in increasing function and in decreasing pain related to RCT. However, the lack of studies comparing different types of exercises (i.e. concentric, eccentric, scapular strengthening, proprioceptive, coactivation) is reported by many systematic reviews. One type of exercise, coactivation strengthening, could be more efficient. Coactivation strengthening implies a recruitment of the pectoralis major and the latissimus dorsi while performing regular strengthening. When theses muscles are recruited, the medio-inferior orientation of their tendons creates a force vector that limits the superior translation of the humeral head, thus limits the subacromial narrowing.

The aim of this study is to evaluate the efficacy of coactivation strengthening exercises in patient with RCT compared to regular strengthening exercises. Forty-two participants diagnosed with RCT by an orthopaedic surgeon following a standardized protocol will be randomised to either coactivation or regular strengthening exercises. Participants will perform a 6-week exercise protocols. Outcomes will be measured at baseline, and at three, six, 12, 18 and 24 weeks. The primary outcome is function assessed with the Disabilities of arm, shoulder and Hand (DASH) questionnaire. Secondary outcomes focus on pain (visual analog scale), quality of life (Western Ontario Rotator Cuff Index), impression of change (Patient Global Impression of Change), subacromial distance (ultrasonography) and muscular strength (manual dynamometer). Investigators expect that coactivation strengthening exercises will be more efficient over the short and long term.

This trial will provide data to guide clinicians in the treatment of RCT to reduce recovery time and to bring patients back as quickly as possible to work or usual function.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Experienced shoulder pain > four weeks
* Positive Painful Arc Test
* Positive Neer or Hawkins Kennedy test
* Pain at resisted isometric movement of abduction or external rotation

Exclusion Criteria:

* Any other shoulder pathology
* Rotator cuff complete tear
* History of shoulder surgery
* Any systemic inflammation or neurological condition
* Received a corticosteroid injection < six weeks
* Any known cognitive condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-07; Primary Completion 2017-10 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Change in function (Disabilities of Arm, Shoulder and Hand Questionnaire - DASH) | Baseline - six weeks
  DASH is a self-reported questionnaire of 30 items measuring physical disability and symptoms. (St-Pierre et al., 2015; Roy et al., 2009)

SECONDARY OUTCOMES:
Change in function (Disabilities of Arm, Shoulder and Hand Questionnaire - DASH) | Baseline - three, 12, 18 and 24 weeks
  DASH is a self-reported questionnaire of 30 items measuring physical disability and symptoms. (St-Pierre et al., 2015; Roy et al., 2009)
Change in pain (Visual Analogue Scale - VAS) | Baseline - three, six, 12, 18 and 24 weeks
  VAS is a self-reported scale of 10 cm measuring the intensity of pain from 0 (no pain) to 10 cm (worst pain). (Dworkin et al., 2008)
Change in quality of life/Function (Western Ontario Rotator Cuff Index - WORC) | Baseline - three, six, 12, 18 and 24 weeks
  WORC index is a disease-specific questionnaire developed to measure health related quality-of-life of individuals suffering from RC disorders. It contains 21 items divided into five sections: physical symptoms, sports/recreation, work, lifestyle and emotions. (Ekeberg et al., 2010)
Impression of Change (Patient Global Impression of Change - PGIC) | at three, six, 12, 18 and 24 weeks
  PGIC is a single-item rating by participants of their response during a clinical trial using a seven-points rating scale between "Very much worst" and "Very much improved". (Dworkin et al., 2008)
Change in subacromial distance (ultrasound scanner) | Baseline - six weeks
  Subacromial distance is defined as the tangential distance between the upper part of the humeral head and the lower part of the acromion. Ultrasound Imaging will be performed with a 6-13 Hz linear array probe (Sonosite Turbo, Futjifilm). (Desmeules et al., 2004)
Isometric strength (manual dynamometer) | Baseline - six weeks
  The isometric strength of flexion, abduction, internal and external rotation movements will be perform with a MicroFET manual dynamometer (Hoggan Health Industries, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Nathaly Gaudreault, Ph.D., Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de Recherche du CHUS, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ostor AJ, Richards CA, Prevost AT, Speed CA, Hazleman BL. Diagnosis and relation to general health of shoulder disorders presenting to primary care. Rheumatology (Oxford). 2005 Jun;44(6):800-5. doi: 10.1093/rheumatology/keh598. Epub 2005 Mar 15. PMID 15769790
- [Background] Papadonikolakis A, McKenna M, Warme W, Martin BI, Matsen FA 3rd. Published evidence relevant to the diagnosis of impingement syndrome of the shoulder. J Bone Joint Surg Am. 2011 Oct 5;93(19):1827-32. doi: 10.2106/JBJS.J.01748. PMID 22005869
- [Background] MacDermid JC, Ramos J, Drosdowech D, Faber K, Patterson S. The impact of rotator cuff pathology on isometric and isokinetic strength, function, and quality of life. J Shoulder Elbow Surg. 2004 Nov-Dec;13(6):593-8. doi: 10.1016/j.jse.2004.03.009. PMID 15570226
- [Background] Graichen H, Hinterwimmer S, von Eisenhart-Rothe R, Vogl T, Englmeier KH, Eckstein F. Effect of abducting and adducting muscle activity on glenohumeral translation, scapular kinematics and subacromial space width in vivo. J Biomech. 2005 Apr;38(4):755-60. doi: 10.1016/j.jbiomech.2004.05.020. PMID 15713296
- [Background] Hanratty CE, McVeigh JG, Kerr DP, Basford JR, Finch MB, Pendleton A, Sim J. The effectiveness of physiotherapy exercises in subacromial impingement syndrome: a systematic review and meta-analysis. Semin Arthritis Rheum. 2012 Dec;42(3):297-316. doi: 10.1016/j.semarthrit.2012.03.015. Epub 2012 May 18. PMID 22607807
- [Background] Beaudreuil J, Lasbleiz S, Aout M, Vicaut E, Yelnik A, Bardin T, Orcel P. Effect of dynamic humeral centring (DHC) treatment on painful active elevation of the arm in subacromial impingement syndrome. Secondary analysis of data from an RCT. Br J Sports Med. 2015 Mar;49(5):343-6. doi: 10.1136/bjsports-2012-091996. Epub 2013 Mar 23. PMID 23525552
- [Background] St-Pierre C, Dionne CE, Desmeules F, Roy JS. Reliability, validity, and responsiveness of a Canadian French adaptation of the Western Ontario Rotator Cuff (WORC) index. J Hand Ther. 2015 Jul-Sep;28(3):292-8; quiz 299. doi: 10.1016/j.jht.2015.02.001. Epub 2015 Feb 14. PMID 25990445
- [Background] Roy JS, MacDermid JC, Woodhouse LJ. Measuring shoulder function: a systematic review of four questionnaires. Arthritis Rheum. 2009 May 15;61(5):623-32. doi: 10.1002/art.24396. PMID 19405008
- [Background] Dworkin RH, Turk DC, Wyrwich KW, Beaton D, Cleeland CS, Farrar JT, Haythornthwaite JA, Jensen MP, Kerns RD, Ader DN, Brandenburg N, Burke LB, Cella D, Chandler J, Cowan P, Dimitrova R, Dionne R, Hertz S, Jadad AR, Katz NP, Kehlet H, Kramer LD, Manning DC, McCormick C, McDermott MP, McQuay HJ, Patel S, Porter L, Quessy S, Rappaport BA, Rauschkolb C, Revicki DA, Rothman M, Schmader KE, Stacey BR, Stauffer JW, von Stein T, White RE, Witter J, Zavisic S. Interpreting the clinical importance of treatment outcomes in chronic pain clinical trials: IMMPACT recommendations. J Pain. 2008 Feb;9(2):105-21. doi: 10.1016/j.jpain.2007.09.005. Epub 2007 Dec 11. PMID 18055266
- [Background] Ekeberg OM, Bautz-Holter E, Keller A, Tveita EK, Juel NG, Brox JI. A questionnaire found disease-specific WORC index is not more responsive than SPADI and OSS in rotator cuff disease. J Clin Epidemiol. 2010 May;63(5):575-84. doi: 10.1016/j.jclinepi.2009.07.012. PMID 19836206
- [Background] Desmeules F, Minville L, Riederer B, Cote CH, Fremont P. Acromio-humeral distance variation measured by ultrasonography and its association with the outcome of rehabilitation for shoulder impingement syndrome. Clin J Sport Med. 2004 Jul;14(4):197-205. doi: 10.1097/00042752-200407000-00002. PMID 15273525
- [Derived] Boudreau N, Gaudreault N, Roy JS, Bedard S, Balg F. The Addition of Glenohumeral Adductor Coactivation to a Rotator Cuff Exercise Program for Rotator Cuff Tendinopathy: A Single-Blind Randomized Controlled Trial. J Orthop Sports Phys Ther. 2019 Mar;49(3):126-135. doi: 10.2519/jospt.2019.8240. Epub 2018 Nov 30. PMID 30501388